CLINICAL TRIAL: NCT00318006
Title: A Randomized Study of Nasal Irrigation Versus Nasal Spray for Chronic Nasal and Sinus Symptoms
Brief Title: Study of Nasal Irrigation Versus Nasal Spray for Chronic Nasal and Sinus Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: NeilMed Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Melissa Pynnonen, Associate Professor of Otolaryngology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HUM00000253
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Rhinosinusitis
Keywords: chronic; nasal; sinus; symptoms
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Fistula

ARMS (2):
- Spray (Active Comparator): subjects were instructed in the technique of nasal lavage (irrigation group) or nasal saline spray (spray group) and were asked to do the assigned treatment twice daily for 8 weeks. They were provided with an 8-week supply of materials (Sinus Rinse irrigations from NeilMed Products Inc, and Deep Sea nasal saline spray distributed by Major Pharmaceuticals, Livonia, Michigan).
  Interventions: Procedure: saline spray
- Irrigation (Experimental): subjects were instructed in the technique of nasal lavage (irrigation group) or nasal saline spray (spray group) and were asked to do the assigned treatment twice daily for 8 weeks. They were provided with an 8-week supply of materials (Sinus Rinse irrigations from NeilMed Products Inc, and Deep Sea nasal saline spray distributed by Major Pharmaceuticals, Livonia, Michigan).
  Interventions: Procedure: saline irrigation

INTERVENTIONS:
Procedure: saline irrigation — subjects were instructed in the technique of nasal lavage (irrigation group) or nasal saline spray (spray group) and were asked to do the assigned treatment twice daily for 8 weeks. They were provided with an 8-week supply of materials (Sinus Rinse irrigations from NeilMed Products Inc, and Deep Sea nasal saline spray distributed by Major Pharmaceuticals, Livonia, Michigan).
  Arms: Irrigation
Procedure: saline spray — subjects were instructed in the technique of nasal lavage (irrigation group) or nasal saline spray (spray group) and were asked to do the assigned treatment twice daily for 8 weeks. They were provided with an 8-week supply of materials (Sinus Rinse irrigations from NeilMed Products Inc, and Deep Sea nasal saline spray distributed by Major Pharmaceuticals, Livonia, Michigan).
  Arms: Spray

SUMMARY:
This study will compare nasal saline irrigation with nasal saline spray for the treatment of chronic nasal and sinus symptoms. Participants will complete a questionnaire regarding their nasal and sinus symptoms and will be randomly assigned to one of the treatment groups. Each participant will be instructed on how to perform daily nasal treatment.The subjects will complete follow-up surveys at regular intervals to assess any change in their nasal symptoms after starting nasal saline treatment. Participants may take their usual medications for sinus symptoms during their participation in the study.

DETAILED DESCRIPTION:
See publication: Arch OtolaryngolHeadNeckSurg. 2007;133(11):1115-1120

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Presence of any one of the following symptoms for > 4 days/week and > 15 days in the past 1 month:

  * Nasal stuffiness
  * Nasal congestion
  * Nasal dryness or crusting
  * Abnormal nasal discharge
  * Thick nasal discharge

Exclusion Criteria:

* Functional endoscopic sinus surgery (FESS) in the last 3 months
* Epistaxis in the last 3 months that required treatment
* Acute illness like otitis media, laryngitis, pharyngitis, or rhinitis in the last 2 weeks
* Acute attack of asthma or bronchitis in the last 2 weeks
* Inability to speak or read English
* Current use of any of the study medications regularly for more than a week in the last 1 month
* Any history of intolerance to saline treatment (if used)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2005-12; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change in the mean score of the sinonasal outcome test-20
Change in medication usage for nasal and sinus symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Pynnonen, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Pynnonen MA, Mukerji SS, Kim HM, Adams ME, Terrell JE. Nasal saline for chronic sinonasal symptoms: a randomized controlled trial. Arch Otolaryngol Head Neck Surg. 2007 Nov;133(11):1115-20. doi: 10.1001/archotol.133.11.1115. PMID 18025315
- See also: Related Info — http://www.umms.med.umich.edu